CLINICAL TRIAL: NCT00158028
Title: Risperidone in the Treatment of Psychotic-like and Deficit Symptoms of Schizotypal Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Harold W Koenigsberg, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 94-561
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Schizotypal Personality Disorder
Keywords: Schizotypal Personality Disorder; Risperidone; Treatment; Cognitive
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone (Experimental): starting dose 0.25mg/day, titrated upward to 2mg/day over 9 weeks
  Interventions: Drug: Risperidone
- Placebo (Placebo Comparator): placebo match in identical tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — The dosage of risperidone was titrated upward in a stepwise design, beginning with 0.25 mg/d for the first week, 0.5 mg/d for weeks 2 and 3, 1.0 mg/d for weeks 4 and 5, 1.5 mg/d for weeks 6 and 7, and 2.0 mg/d for the remaining weeks.
  Arms: Risperidone
Drug: Placebo — placebo match in identical tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of risperidone compared to placebo in the treatment of the psychotic-like and deficit symptoms of schizotypal personality disorder (SPD). Treatment with risperidone, a 5HT2 and dopamine D2 blocking agent, holds particular promise in the treatment of SPD. Unlike traditional antipsychotics, risperidone targets the deficit or negative symptoms of schizophrenia. The deficit-like symptoms of SPD are therefore also likely respond to treatment with risperidone. One common complication in the present psychopharmacologic treatment of SPD with traditional neuroleptics is the fact that many patients discontinue treatment due to the medication-induced dysphoria. Given initial reports and the serotonergic component of the risperidone mechanism, risperidone is anticipated to produce little or no dysphoria.

DETAILED DESCRIPTION:
All patients receive a comprehensive medical evaluation prior to their participation in any studies, as part of their normal clinical care. The evaluation includes an extensive medical history, physical examination, and laboratory evaluation including SMA-18, CBC with differential, TFT's, U/A, stool guaiac, serology, drug screen, chest X-ray (where indicated), EKG, and, for women, pregnancy test. [Note: Subjects will have consented to these procedures in a separate consent, "Biological Correlates of Personality Disorder- Information for Subjects (88244)", before being invited to join this study.] Patients will be interviewed by clinical psychology doctoral students trained in the use of structured instruments to assess Axis I and Axis II pathology. A rater will independently complete either the Schedule for Affective Disorders and Schizophrenia (SADS) (Spitzer & Endicott 1978), modified for evaluation of DSM-IV criteria for Axis 1 disorders, or the Structured Clinical Interview for DSM-IV Axis I Disorders ( First et al 1996) and the Structured Interview for DSM-III-R Personality Disorders (SIDP-R) (Pfohl et al 1989) also modified for the evaluation of DSM-IV criteria. When possible, information will be gathered independently from an informant (first degree relative or life-long friend) to supplement information obtained from clinical interviews and review of past records. The use of structured interviews, and questionnaires are not part of standard clinical care.

PART 1 Part 1 is a single-blind two-week placebo washout. Patients will be seen weekly by a research psychiatrist. One week of (placebo) medication will be dispensed at a time by a research program physician under the direct supervision of Dr. Koenigsberg. Patients will be seen weekly throughout the study. Interviews and assessments are standardized and identical throughout all phases of the study. They include the Clinical Global Impression scale (CGI), the Scale for the Assessment of Negative Symptoms (SANS), the Positive and Negative Symptom Scale (PANSS), and the Hamilton Depression Rating Scale (HDRS), all administered weekly. At baseline and after 4- and 9-weeks of treatment, subjects will also receive a series of paper-and-pencil and computer-presented cognitive tests (DOT test, Paced Auditory Serial Addition Task, Continuous Performance Task-Identical Pairs version, Serial Verbal Learning Test and the Wechsler memory Scale-Revised Visual Reproduction test). No medications, other than study drug, are allowed during the protocol. If, during this two-week placebo washout period, the total SANS score decreases by 35% or greater, patients will not be entered into Phase 2. Use of a placebo washout is not part of standard clinical care.

PART 2 Part 2 is the double blind, 9-week parallel-arm placebo-controlled portion of the study. Randomization will be conducted by the Pharmacy. One week of medication (active or placebo) will be dispensed at a time by a research program physician under the direct supervision of Dr. Koenigsberg. The patient will receive 1 tablet PO QD every day of the study. If enrolled in the Active Arm of the study, the patient will receive a .25 mg risperidone tablet orally once daily for Days 1 to 7; .5 mg risperidone tablet orally once daily for Days 8 to 21; 1 mg risperidone tablet orally once daily for Days 22-35; 1.5 mg risperidone tablet orally once daily for days 36-49; and a 2 mgs of risperidone orally once daily for days 50 to 63. If the treating psychiatrist believes that a higher dose is clinically indicated, the physician may alter the above by increasing the dose to 2 mg per day beginning on day 22 and to 4 mg per day beginning on day 50. Weekly visits will include standard assessment and review of protocol compliance. Treatment with risperidone is not part of current standard clinical care of schizotypal personality disorder and this study is designed to establish its usefulness with this population. Similarly use of a double bind placebo control is not part of standard clinical care.

PART 3 Patients who were randomized into the placebo arm of Part 2 will be offered the opportunity of participating in an 8 week open label study of risperidone otherwise identical to Part 2.

Data will be analyzed by a repeated measures analysis of variance separately for scores on the CGI, SANS, PANSS, and HDSR comparing placebo and active medication.

ELIGIBILITY:
Inclusion Criteria:

Schizotypal Personality Disorder

Exclusion Criteria:

Over 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1995-11; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANAS) rating

SECONDARY OUTCOMES:
Clinical global Impression, Schizotypal Persoality Questionarre Score, CPT-IP, Paced Auditory Serial Addition Task, Wechsler memory scale-Revised Visual Reproduction; Serial Verbal Learning Test

CONTACTS AND LOCATIONS:
Overall Officials: Harold Koenigsberg, Principal Investigator — Mount Sinai School of Medicine/Bronx VA
Locations (1):
- Bronx VA, The Bronx, New York, United States

REFERENCES:
- [Result] Koenigsberg HW, Reynolds D, Goodman M, New AS, Mitropoulou V, Trestman RL, Silverman J, Siever LJ. Risperidone in the treatment of schizotypal personality disorder. J Clin Psychiatry. 2003 Jun;64(6):628-34. doi: 10.4088/jcp.v64n0602. PMID 12823075